CLINICAL TRIAL: NCT04783142
Title: The Influence of Diet on Host Physiology and Disease Across Diverse Human Gut Microbiotas
Brief Title: A Study to Evaluate the Influence of Diet on GI Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Purna C. Kashyap, MBBS, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20-008067
Record Dates: First submitted 2021-02-23; First posted 2021-03-05 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: High-Protein, Low-Fiber Diet
MeSH Terms: interventions — Diet, Protein-Restricted; Diet, High-Protein

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the high-fiber, low protein diet or the low-fiber, high-protein diet.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Principal investigator and analysts will be blinded. The participant will not be told to which diet they are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fiber, low-protein diet (Other): Participants will consume a high-fiber, low-protein diet for at least 4 weeks. All meals will be provided free of charge. No substitutions will be permitted.
  Interventions: Other: High-fiber, low-protein diet
- Low-fiber, high-protein diet (Other): Participants will consume a low-fiber, high-protein diet for at least 4 weeks. All meals will be provided free of charge. No substitutions will be permitted.
  Interventions: Other: Low-fiber, high-protein diet

INTERVENTIONS:
Other: High-fiber, low-protein diet — Diet will consist of at least 15g fiber above baseline and less than 10% of calories from protein.
  Arms: High-fiber, low-protein diet
Other: Low-fiber, high-protein diet — Diet will consist of less than 15g fiber and greater than 18% of calories from protein
  Arms: Low-fiber, high-protein diet

SUMMARY:
The purpose of this study is to understand the potential of protein and psyllium fiber to manipulate gut microbial densities, intestinal permeability, and inflammation in humans.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* On a baseline diet characterized by: Fiber intake of </= 20g/day, > 18% of daily calories from protein

Exclusion Criteria:

* Prior history of gastrointestinal surgeries (except appendectomy and cholecystectomy)
* Known diagnosis of inflammatory bowel disease (Crohn's or ulcerative colitis), microscopic colitis, celiac disease, or other inflammatory GI condition
* Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability)
* Use of NSAIDs or aspirin and unable or unwilling to stop taking two weeks prior to permeability test and for the duration of the study
* Use of osmotic laxatives and unable or unwilling to stop taking one week prior to permeability test and for the duration of the study
* Use of oral corticosteroids and unable or unwilling to stop use of oral corticosteroids within the previous 6 weeks and for the duration of the study
* Multiple dietary restrictions or unable/unwilling to alter dietary protein or dietary fiber.
* Unwilling to stop ingestion of alcohol and artificial sweeteners such as Splenda™ (sucralose), Nutrasweet™ (aspartame), sorbitol, xylitol, lactulose, or mannitol 2 days before and during the permeability testing days, e.g. foods to be avoided are sugarless gums or mints and diet beverages
* Unwilling to stop stenuous exercise (running >5 miles or equivalent) one week prior to the permeability tests
* Bowel preparation for colonoscopy less than one week prior to completion of the first stool kit and permeability test and flexible sigmoidoscopy and upper endoscopy
* Pregnancy or plan to become pregnant during the study time frame
* Vulnerable adult
* Known bleeding disorders or takes medications that increase risk of bleeding from mucosal biopsies
* Use of oral antibiotic(s) within the past 4 weeks (can be enrolled after 4-week washout period)
* Use of commercial probiotic formulations and unwilling to stop for the duration of the study
* Diagnosis of diabetes
* Any other disease(s), condition(s) or habits(s) that would interfere with completion of study, or in the judgment of the investigator would potentially interfere with compliance to this study or would adversely affect study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-03-27 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of Lactulose and 13C-Mannitol | 4 weeks
  Small Bowel and Colonic Permeability by Urinary Excretion of Lactulose and 13C-Mannitol after Oral Ingestion of lactulose and 13C mannitol (5:1 ratio by mass). The 0-2h urine most closely reflects small intestinal permeability and 8-24h urine reflects colonic permeability. HPLC-tandem mass spectrometry will be used for detection of the sugars. The results will be expressed as the ratio of percentage excretion of the ingested dose of lactulose and mannitol in urine.

SECONDARY OUTCOMES:
Change in gut microbial alpha diversity based on Shannon index | 4 weeks
  Stool samples will be processed to extract DNA, followed by metagenomic sequencing and assessment of alpha diversity using Shannon index. Comparison will be made using ttest.

CONTACTS AND LOCATIONS:
Overall Officials: Purna C. Kashyap, MBBS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials